CLINICAL TRIAL: NCT02675153
Title: Efficacy and Safety of Rapamycin in the Treatment of Crohn's Disease-related Stricture
Brief Title: To Evaluate the Efficacy and Safety of Rapamycin for Crohn's Disease-related Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Associate professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPA-CN-160122
Record Dates: First submitted 2016-01-21; First posted 2016-02-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Crohn's Diseases
Keywords: rapamycin; stricture; fibrosis
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic; Fibrosis | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Upper gastrointestinal strictures (Experimental): Patients with upper gastrointestinal strictures were treated with rapamycin (2mg/day, Sirolimus, Roche) for at least six months.
  Interventions: Drug: Rapamycin
- Lower gastrointestinal strictures (Experimental): Patients with lower gastrointestinal strictures were treated with rapamycin (2mg/day, Sirolimus, Roche) for at least six months.
  Interventions: Drug: Rapamycin

INTERVENTIONS:
Drug: Rapamycin — Participants with gastrointestinal strictures were treated with rapamycin 2mg daily at least six months.
  Other Names: Sirolimus

SUMMARY:
Crohn's disease （CD） with stenosis has limited therapeutic options and with high surgical rate. The present clinical trial aims to evaluate the efficacy and safety of rapamycin in the treatment of stricturing Crohn's Disease.

DETAILED DESCRIPTION:
Management of Crohn's disease （CD） with stenosis is challenging and often requires endoscopic dilatation or surgical resection of the strictured bowel. Sirolimus (rapamycin), a macrocyclic antibiotic with immunosuppressive and antineoplastic properties, has been reported as promising rescue therapy for refractory CD. This study aims to evaluate the use of sirolimus for stricturing Crohn's Disease. Patients in this study will receive a continuous dosing schedule of oral sirolimus 2mg daily for six months. Clinical responses were defined as the ability to tolerate the regular diet with vegetable fiber combined with a reduction of ≥ 75% in overall target score and a score of less than two points for each item.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese patients (≥18 years of age) with a documented definite diagnosis of CD;
2. the presence of a clinically symptomatic stricture;
3. strictures confirmed by endoscopy (passage of the endoscope with resistance or not traversable) or imaging (CT enterography (CTE) or MR enterography (MRE).

Exclusion Criteria:

1. Patients who were pregnant, diagnosed with intestinal perforation, complete intestinal obstruction, any signs of dysplasia or malignancy, or use of anti-tumor necrosis factor (TNF) in the last three months;
2. Patients who were not followed up between the inception of medication and any other subsequent treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Response rate | up to 24 weeks
  Response was defined as the following criteria: (a) the ability to tolerate a normal diet (vegetable fiber), with a reduction of ≥ 75% in overall baseline target score and sub-score ≤ 2 (Table S1); (b) no need for ED or surgery; (c) no severe adverse events or any other reasons leading to rapamycin withdrawal.

SECONDARY OUTCOMES:
Adverse events | through study completion, an average of 3 years
  New onset of symptoms and the exacerbation of previous symptoms were recorded as adverse events (AEs)
The rate of surgery or ED after rapamycin | through study completion, an average of 3 years
  For long-term treatment outcomes, the primary endpoint was the rate of surgery or ED after rapamycin.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, MD,PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Mutalib M, Borrelli O, Blackstock S, Kiparissi F, Elawad M, Shah N, Lindley K. The use of sirolimus (rapamycin) in the management of refractory inflammatory bowel disease in children. J Crohns Colitis. 2014 Dec;8(12):1730-4. doi: 10.1016/j.crohns.2014.08.014. Epub 2014 Sep 18. PMID 25240477
- [Background] Massey DC, Bredin F, Parkes M. Use of sirolimus (rapamycin) to treat refractory Crohn's disease. Gut. 2008 Sep;57(9):1294-6. doi: 10.1136/gut.2008.157297. PMID 18719139